CLINICAL TRIAL: NCT01603238
Title: An Open Label, Single-Dose, Study in Healthy Male Subjects Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C] LC15-0444
Brief Title: Study in Healthy Male Subjects Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C] LC15-0444
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL008
Record Dates: First submitted 2012-05-17; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Healthy

ARMS (1):
- [14C]-LC15-0444 (Experimental): A single oral dose of [14C]-LC15-0444 50 mg , containing 4.9 MBq [14C] (batch number 110372/C/01).
  Interventions: Drug: [14C]-LC15-0444

INTERVENTIONS:
Drug: [14C]-LC15-0444 — A single oral administration of [14C]-LC15-0444 50 mg, containing 4.9 MBq [14C]. Subjects in the fasted state will receive the drug as a capsule, with 240 ml of water.

SUMMARY:
This was an open-label, non-randomised, single-dose study in 6 healthy male subjects. Subjects attended a screening visit within 28 days before drug administration. Subjects were admitted to the clinical unit on the morning of the day before dosing (Day -1) and received a single oral administration of study drug in a fasted state on Day 1. Subjects were resident in the clinic for up to 7 days after dosing; they could be discharged sooner if a mass balance cumulative recovery of >95% was achieved, or if a mass balance cumulative recovery of >90% was achieved and <1% was collected within 2 separate, consecutive 24 h periods. At specified times during the study period, blood samples were taken and urine and faeces were collected for PK analysis. Safety assessments were also performed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 30 to 65
2. Body Mass Index (BMI) of 18-35 kg/m2
3. Must be willing and able to communicate and participate in the whole study
4. Must provide written informed consent
5. Subject must agree to use an adequate method of contraception, during the study and for 12 weeks after the last dose of the investigational drug. Male subjects will be instructed to use appropriate contraception, including a barrier method (condom), in addition to any precautions taken by their partner;
6. Normal (or abnormal but not clinically significant) supine blood pressure (BP) and heart rate (HR)
7. Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment (detailed medical history and a complete physical examination),electrocardiogram (ECG) and laboratory investigations (haematology, blood chemistry and urinalysis).

Exclusion Criteria:

1. Participation in a clinical research study involving investigational drugs or dosage forms within the previous 3 months
2. Subjects who have previously been enrolled in this study
3. History of any drug or alcohol abuse in the past 2 years
4. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine);
5. Subjects who admit to any current or previous use of Class A drugs such as opiates, cocaine, ecstasy, lysergic acid diethylamide (LSD) and intravenous amphetamines (Subjects who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs of abuse test and have been abstinent for at least 12 months)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at admission
7. Radiation exposure from clinical studies, including that from the present study,excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last twelve months or 10 mSv in the last five years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 72h post dose
  Whole blood and plasma concentrations of total radioactivity

SECONDARY OUTCOMES:
Cmax | up to 72h post dose
  Plasma concentrations of parent drug

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair MBChB, Principal Investigator — Quotient Bioresearch Clinical Services
Locations (1):
- LG Life Sciences, Seoul, South Korea